CLINICAL TRIAL: NCT06994078
Title: Clinical Application of PET Imaging Targeting Nectin-4 in Malignant Tumors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XLan-0519
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Urothelial Carcinoma; Breast Cancer; Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell; Breast Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET imaging targeting Nectin-4 in malignant tumors (Experimental): Determine if targeting Nectin-4 PET is safe and effective method for imaging of malignant tumors.
  Interventions: Drug: 68Ga-NOTA-Nectin-4 antibody fragment

INTERVENTIONS:
Drug: 68Ga-NOTA-Nectin-4 antibody fragment — To perform integrated PET/MR or PET/CT visualization of patients with clinically suspected or confirmed urothelial carcinoma, breast cancer, lung carcinoma and other malignant tumors with high Nectin-4 expression and healthy volunteers, using specific positron imaging agents targeting Nectin-4 (taking [68Ga]Ga-NOTA-Nectin-4 antibody fragment as an example), to achieve the following purposes: Patients with malignant tumors: for diagnosis and staging of diseases, comparing with the gold standard pathological diagnosis, evaluating diagnostic efficacy, clarifying the presence or absence of lesions, and determining the location and nature of lesions; comparing with [18F]FDG PET for accurate staging, evaluating the tumor load, and helping to determine the therapeutic plan. Healthy volunteers: Pharmacokinetic analysis will be performed to clarify the distribution and metabolism of the drug in the body and its safety.

SUMMARY:
This study is a diagnostic study. Patients and healthy volunteers with clinically suspected or confirmed urothelial carcinoma, breast cancer, lung carcinoma and other malignant tumors with high expression of Nectin-4 will be recruited for PET/MR or PET/CT imaging targeting a Nectin-4-specific probe (in the case of [68Ga]Ga-NOTA-Nectin-4 antibody fragment) , to observe the reaction of volunteers and patients after injection of drugs, to evaluate the pharmacokinetics in vivo and the efficacy of diagnosis and staging, and to perform PET imaging in patients with contraindications. General information on the subjects' vital signs, clinical data, blood routine, liver and kidney functions and other biochemical indicators and other imaging data were collected, and histopathology of biopsy or surgical specimens was used as the final diagnostic criterion.

DETAILED DESCRIPTION:
Malignant tumors are one of the major diseases leading to death worldwide, and their high incidence and mortality rates pose a serious threat to human health. According to the World Health Organization (WHO), there will be about 19.3 million new cancer cases and 10 million deaths globally in 2020, with a significant increase in the incidence of malignant tumors such as lung and breast cancers in particular. Early diagnosis and load assessment of tumors are crucial for improving patient survival.

Currently, there are limitations in the commonly used clinical diagnostic imaging tools. For example, traditional anatomical imaging techniques (e.g., ultrasound, CT, and MRI) have high resolution in displaying the anatomical structure of tumors, but it is difficult to accurately differentiate between benign and malignant lesions, and is not sufficiently sensitive to the performance of some tumors rich in fibrotic and necrotic tissues. Enhanced magnetic resonance imaging (ceMRI) has limited effectiveness in the detection of certain solid tumors, and is particularly deficient in the identification of microscopic lesions and some deep tumors. [18F]FDG PET/CT, a current widely used molecular imaging technique, enables functional imaging of tumors by reflecting the level of glucose metabolism. However, [18F]FDG is not a tumor-specific imaging agent, and non-malignant lesions such as inflammation, infection, and tuberculosis can also lead to an increase in local FDG uptake, producing false-positive results. In addition, [18F]FDG uptake is low in some tumors with low metabolic activity (e.g., poorly differentiated carcinomas and some brain tumors), leading to false-negative results and limiting its use in early tumor diagnosis and precision assessment. Therefore, the development of more specific and sensitive molecular imaging probes has significant clinical value.

Nectin-4, a cell adhesion molecule, belongs to an important member of the Nectin family, which is mainly expressed in the embryonic developmental stage and is less expressed in normal adult tissues. However, studies have shown that Nectin-4 is highly expressed in a variety of malignant tumors, including bladder, breast, lung, ovarian and pancreatic cancers, etc. It is closely related to tumor proliferation, invasion, metastasis, and the poor prognosis of patients, and it has gradually become a potential marker for tumor diagnosis and treatment. Especially in bladder cancer, the high expression of Nectin-4 is closely related to tumor stage and malignancy degree, and has become an important molecular target for targeted therapy. In recent years, breakthroughs have been made in the research of targeted drugs against Nectin-4, and the U.S. FDA has approved Enfortumab Vedotin (EV), the first antibody-drug coupling (ADC) targeting Nectin-4, for the treatment of recurrent or refractory uroepithelial cancers, which has shown remarkable efficacy and good prospects for clinical application. However, how to screen patients suitable for targeted Nectin-4 therapy and dynamically evaluate the therapeutic efficacy remain clinical challenges. Therefore, the development of molecular imaging probes targeting Nectin-4 and the realization of non-invasive, real-time quantitative detection of Nectin-4 expression by PET imaging are expected to provide an imaging basis for targeted therapy. This can not only be used to screen patient groups with high Nectin-4 expression, thus precisely guiding the clinical application of targeted drugs, but also to assess drug efficacy in real time during the treatment process and promote the implementation of individualized treatment plans.

In summary, the aim of this project is to explore the clinical application of PET imaging technology targeting Nectin-4 in malignant tumors, through the use of targeted Nectin-4 PET imaging agent (in the case of [68Ga]Ga-NOTA-Nectin-4 antibody fragment) with a view to be used for diagnosis and staging of malignant tumor patients, assessing tumor load and Nectin-4 expression abundance, and helping to determine therapeutic options. At the same time, preliminary pharmacokinetic analysis was performed in healthy volunteers to clarify the metabolic pattern and adverse effects of the drug in vivo.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet all enrollment criteria to be eligible to participate in the study:

* 1: The subject or his/her legal representative is able to sign and date the informed consent form;
* 2: A commitment to comply with the research procedures and to cooperate in the implementation of the full research process;
* 3: Adult patients or healthy volunteers (aged 18 or above) of either sex;
* 4: Patients with clinically suspected or confirmed malignant tumors such as urothelial carcinoma, breast cancer and lung carcinoma (supporting evidence includes serum-related tumor markers, imaging data such as ultrasound, CT, MRI, etc., and histological pathology examination, etc.) and in good general condition;
* 5: Consistent with the results of specific laboratory tests;
* 6: Females of childbearing potential who have been using contraception for at least one month prior to screening and who are committed to using contraception for the entire study period and until a specified time after the end of the study；
* 7: Other set entry criteria.

Exclusion Criteria:

All subjects who meet any of the exclusion criteria baseline will be excluded from the study:

* 1: Those who are unable to complete a PET/MR or PET/CT examination (including inability to lie down, claustrophobia, radiophobia, etc.);
* 2: Having other comorbidities;
* 3: Patients with known hypersensitivity to Nectin-4 antibody fragment developers or synthetic excipients; fasting blood glucose level greater than 11.0 mmol/L prior to 18F-FDG injection；
* 4: Have a history of comorbid drug use;
* 5: Patients considered by the investigator to have poor compliance;
* 6: Patients during pregnancy or lactation;
* 7: Persons with other factors that make participation in this test inappropriate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Visual and standardized uptake values assessment of lesions and biodistribution | 1 year
  At least two experienced nuclear medicine physicians will conduct a visual analysis using consensus reading. The standardized uptake value (SUV) of tumor and organs will be measured after a semiquantitative analysis is conducted for each case. The SUV ranges from 0 to infinity, and a higher score means a higher uptake of targeting Nectin-4 nuclear probe by the tumor, which implies a greater threat of the tumor being malignant or higher stage.

SECONDARY OUTCOMES:
Radioactivity in the blood and urine samples | 1 year
  Blood samples were collected at 25 minutes, 55 minutes and 115 minutes after injection.
Pathological sections of tumour tissue | 1 year
  The excised tumour tissue was taken for immunohistochemistry to verify its Nectin-4 expression

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No